CLINICAL TRIAL: NCT03586635
Title: Automated EDSS Score Calculation Using a Smartphone Application in Multiple Sclerosis Patients
Brief Title: Automated EDSS Score Calculation by Smartphone Application
Acronym: Easy EDSS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 18-PP-09
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: MS CHRONIC PROGRESSIVE

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Multiple Sclerosis
  Interventions: Other: neurological exam

INTERVENTIONS:
Other: neurological exam — Patients participating in the study are recruited from the investigator's tertiary multiple sclerosis management centre. They are systematically examined neurologically as part of their routine follow-up.
  the patient will be exceptionally examined by two distinct persons, a senior doctor and a junior doctor (internal or external) independently.
  At the end of the neurological examination, each examiner will evaluate the EDSS score in a classical way (using paper definitions) then using the smartphone application

SUMMARY:
The EDSS score is the reference tool for rating disability in patients with multiple sclerosis. It is used in both daily monitoring and clinical research studies.

Its main shortcoming lies in its imprecise and variable nature, with significant inter-examiner variability. This variability is the consequence of the complexity of the score rating and also of its subjective nature.

The application developed aims to reduce the risk of rating error, and to homogenize the results obtained regardless of the examiner and his experience in using the score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple sclerosis seen at the Central Nervous System Day Hospital as part of their follow-up and requiring neurological examination.
* Age ≥ 18 years
* No opposition to the use of their data

Exclusion Criteria:

- Neurological or general pathology, other than multiple sclerosis, that may interfere with EDSS score scoring

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - patients coming to the MS Competence and Recovery Centre
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
EDSS score apllication VS paper version | 6 months
  comparison of the overall EDSS score obtained with the application and its paper version at the end of the neurological examination

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No